CLINICAL TRIAL: NCT02184611
Title: A 24 Week Randomised, Double Blind and Placebo Controlled Study to Evaluate the Efficacy and Safety of 62.5 mcg Umeclidinium Inhalation Powder Delivered Once Daily Via a Novel Dry Powder Inhaler in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A 24 Week Efficacy Study of Inhaled Umeclidinium (UMEC) in Patients of Chronic Obstructive Pulmonary Disease (COPD) Using a Novel Dry Powder Inhaler (NDPI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 117410
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: lung function; Umeclidinium; GSK573719; anticholinergic; novel dry powder inhaler; long-acting muscarinic receptor antagonist; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umeclidinium bromide (Experimental): Subjects meeting the eligibility criteria will complete a 7 to 14 day run-in period and will be randomized to receive UMEC Inhalation Powder 62.5 mcg OD over a period of 24 weeks
  Interventions: Drug: Umeclidinium bromide
- Placebo (Placebo Comparator): Subjects meeting the eligibility criteria will complete a 7 to 14 day run-in period and will be randomized to receive matching placebo of UMEC Inhalation Powder OD over a period of 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Umeclidinium bromide — Blended with lactose and magnesium stearate dry white powder of umeclidinium 62.5 mcg to be inhaled via a NDPI
  Arms: Umeclidinium bromide
Drug: Placebo — Blended with lactose and magnesium stearate dry white powder to be inhaled via a NDPI
  Arms: Placebo

SUMMARY:
Studies to date provides substantial evidence for the effectiveness for UMEC 62.5 microgram (mcg) as a long term maintenance therapy for the treatment of COPD; this study further evaluates the efficacy and safety of UMEC 62.5 mcg administered once-daily (OD) for 24 weeks via a NDPI compared with placebo in Asian subjects with COPD. Over approximate 27 weeks of entire study duration, 10 study clinic visits will be conducted on an outpatient basis. Pre-screening visit will be conducted for the informed consent form, review demography, COPD history and COPD concomitant medications. Subjects meeting the eligibility criteria at screening will complete a 7 to 14 day Run-in period and will be provided with albuterol/salbutamol as rescue medication on an "as-needed" basis. Further, subjects will be randomized to the UMEC 62.5 mcg or matching placebo in a 1:2 ratio for 24 week treatment period. A follow up for adverse event assessment will be scheduled approximately 7 days after the treatment period or the Early Withdrawal Visit.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: outpatient, Asian ancestry.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: 40 years of age or older at Screening (Visit 1).
* Gender: Male or female subjects are eligible to participate in the study. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, >45 years, in the absence of hormone replacement therapy. However, in questionable cases, post-menopause status may be confirmed by analysis of a blood sample with follicle-stimulating hormone (FSH) >40 million international units per milliliter (MIU/ml) and estradiol <40 picogram (pg) /ml (<140 picomole per liter (pmol/L) as confirmatory. OR Child bearing potential, provided the subject has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label, and the instructions of the physician for the duration of the study - Screening to Follow-Up contact): Abstinence\ Oral contraceptive either combined or progestogen alone\ Injectable progestogen\ Implants of levonorgestrel\ Estrogenic vaginal ring\ Percutaneous contraceptive patches\ Intrauterine device (IUD) or intrauterine system (IUS)\ Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study and this male is the sole partner for that subject\ Double barrier method condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).
* COPD History: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society as follows: COPD is a preventable and treatable disease state characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
* Tobacco Use and Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >= 10 pack-years [Number of pack years = (number of cigarettes per day /20) x number of years smoked (e.g. 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years both equal 10 pack years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Note: Pipe and/or cigar use cannot be used to calculate pack-year history. COPD patients who only use a pipe and/or cigar are not eligible.
* Severity of Disease: A pre and post-salbutamol/albuterol FEV1/FVC ratio of <0.70 and a pre and post-salbutamol/albuterol FEV1 of <=70% of predicted normal values calculated using National Health and Nutrition Examination Survey III reference equations at Visit 1.
* Dyspnea: A score of >=2 on the Modified Medical Research Council Dyspnoea Scale (mMRC) at Screening (Visit 1)

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis) and lung cancer are absolute exclusionary conditions. A subject, who in the opinion of the investigator has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis or interstitial lung disease.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Chest X-Ray: A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Visit 1 if a chest X-ray or CT scan is not available within 6 months prior to Visit 1.
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* 12-Lead electrocardiogram (ECG): An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1, including the presence of a paced rhythm on a 12-lead ECG which causes the underlying rhythm and ECG to be obscured. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. Specific ECG findings that precluded subject eligibility are as listed. An ECG finding that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following: Sinus tachycardia ≥120 bpm*Note: sinus tachycardia ≥120bpm should be confirmed by two additional readings at least 5 minutes apart. Sinus bradycardia <45bpm*Note: Sinus bradycardia <45bpm should be confirmed by two additional readings at least 5 minutes apart.Multifocal atrial tachycardia.Supraventricular tachycardia (>100bpm).Atrial fibrillation with rapid ventricular response (rate >120bpm). Atrial flutter with rapid ventricular response (rate >120bpm). Ventricular tachycardias (non sustained, sustained, polymorphic, or monomorphic). Ventricular flutter. Ventricular fibrillation. Torsades de Pointes. Evidence of Mobitz type II second degree or third degree atrioventricular (AV) block. AV dissociation. Trifascicular Block. For subjects with QRS duration <120 ms: QTc(F) ≥450msec or an ECG that is unsuitable for QT measurements (e.g., poor defined termination of the T wave). For subjects with QRS duration>120: QTc(F) ≥480msec or an ECG that is unsuitable for QT measurements (e.g., poor defined termination of the T wave). Myocardial infarction (acute or recent) * Note: Evidence of an old (resolved) myocardial infarction is not exclusionary. The study investigator will determine the medical significance of any ECG abnormalities not listed above.
* Screening Labs: Significantly abnormal findings from clinical chemistry and haematology tests at Visit 1.
* Medications Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1 is presented as Medication with Time Interval Prior to Visit 1: Depot corticosteroids (12 weeks); Systemic, oral, parenteral (intra-articular) corticosteroids (4 weeks); Antibiotics (for lower respiratory tract infection) (4 weeks); inhaled corticosteroid/ long-acting beta agonist (ICS/LABA) combination products if ICS/LABA therapy is discontinued completely (30 days); Use of ICS at a dose >1000mcg/day of fluticasone propionate or equivalent (30 days); Initiation or discontinuation of ICS use (30 days); Phosphodiesterase 4 (PDE4) inhibitors (roflumilast) (14 days); Long-acting anticholinergics (e.g.,tiotropium and aclidinium, glycopyronium) (7 days); Theophyllines (12 hours stable dose of theophylline alone is allowed during the study but must be withheld 12 hours prior to each study visit); Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton) (48 hours); Oral beta2-agonists (Long- acting 48 hours, Short -acting 12 hours); Olodaterol and Indacaterol (inhaled long-acting beta2-agonist) (14 days); Salmeterol, formoterol, (inhaled long-acting beta2-agonist) (48 hours); LABA/ ICS combination products only if discontinuing LABA therapy and switching to ICS monotherapy (48 hours for LABA component); Inhaled sodium cromoglycate or nedocromil sodium (24 hours); Inhaled short acting beta2-agonists (4 hours); Inhaled short-acting anticholinergics (e.g. ipratropium bromide) (4 hours, stable dose of ipratropium alone is allowed during the study, provided that the subject is on a stable dose regimen from Screening [Visit 1 and remains so throughout the study] but must be withheld 4 hours prior to each study visit); Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products (4 hours); Any other investigational drug (30 days or 5 half lives, whichever is longer). Note: Further details related to allowable dosage of above listed medications will be explained by the Investigator)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- China (19):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Zhanjiang, Guangdong
  - GSK Investigational Site, Haikou, Hainan
  - GSK Investigational Site, Hohhot, Inner Mongolia
  - GSK Investigational Site, Wuxi, Jiangsu
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Yinchuan, Ningxia
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Qingdao, Shandong
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Shanghai
- South Korea (3):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20367

REFERENCES:
- [Background] Zhong N, Zheng J, Lee SH, Lipson DA, Du X, Wu S. Efficacy and Safety of Once-Daily Inhaled Umeclidinium in Asian Patients with COPD: Results from a Randomized, Placebo-Controlled Study. Int J Chron Obstruct Pulmon Dis. 2020 Apr 17;15:809-819. doi: 10.2147/COPD.S215011. eCollection 2020. PMID 32368027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 09 May 2016 to 08 November 2017 at 26 centers (21 centers in China and 5 centers in the Republic of Korea). A total of 306 participants were included in the Modified Intent-To-Treat (MITT) Population which comprised of all participants randomized to treatment who received at least one dose of study medication.
Pre-assignment Details: Total participants screened were 440; of which, pre-screen failures: 28, Screen failures: 94 (inclusion/exclusion criteria not met: 82, withdrew consent [WC]: 9, adverse event: 2, lost to follow up: 1) and Run in failures: 10 (continuation criteria not met: 6, WC: 4). The remaining 308 participants were randomized (but 2 were randomized in error).
Groups:
- Placebo: Participants received matching placebo to umeclidinium (UMEC) via ELLIPTA® novel dry powder inhaler (DPI) once daily in the morning for the 24-week treatment period.
- UMEC 62.5 mcg: Participants received UMEC 62.5 micrograms (mcg) via ELLIPTA® DPI once daily in the morning for the 24-week treatment period.
Period: Overall Study
Arm/Group | Placebo | UMEC 62.5 mcg
Started | 101 | 205
Completed | 80 | 177
Not Completed | 21 | 28
Not completed — Lack of Efficacy | 11 | 15
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Adverse Event | 4 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Protocol defined stopping criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo to UMEC via ELLIPTA® novel DPI once daily in the morning for the 24-week treatment period.
- UMEC 62.5 mcg: Participants received UMEC 62.5 mcg via ELLIPTA® DPI once daily in the morning for the 24-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC 62.5 mcg | Total
Number analyzed (Participants) | 101 | 205 | 306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (7.05) | 65.5 (6.89) | 65.6 (6.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 16
  Male | 97 | 193 | 290
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 101 | 205 | 306

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough (Pre-bronchodilator) Forced Expiratory Volume in 1 Second (FEV1) on Treatment Day 169
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Treatment Day 169 was defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Treatment Day 168 (i.e. at Week 24). Baseline FEV1 is defined as the mean of the two assessments made pre-dose at Visit 2 (Day 1). Change from Baseline was calculated by subtracting the value on-treatment from the Baseline value. Modified intent-to-treat (mITT) Population comprised of all participants randomized to treatment who received at least one dose of the study medication in the treatment period.
Time Frame: Baseline (Day 1) and Day 169
Population: mITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 80 | 176
Liters | -0.022 (0.0171) | 0.131 (0.0117)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 mcg; UMEC versus Placebo; Test type: Other; p < 0.001, Mixed Models Repeated Measures (MMRM) — Analysis was performed using a MMRM model with covariates of treatment, Baseline, smoking status, country, Day, Day by Baseline and Day by treatment interactions; Least square mean difference = 0.154, 95% CI 2-sided [0.113 to 0.194]

2. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score at Week 24 (Day 168)
Description: The Baseline Dyspnea Index (BDI) is used to measure the severity of dyspnea in participants at Baseline . The TDI measures changes in dyspnea severity from Baseline, as established by the BDI. TDI is formed of 3 individual scales that assess change in functional impairment, change in magnitude of task and change in magnitude of effort. The instrument is scored on a 7-point scale from -3 (major deterioration) to +3 (major improvement) for each category. Total scores (3 categories) range from -9 to +9 with lower scores indicating more deterioration in the severity of dyspnoea. A change of >=1 units is considered to be the minimum clinically important difference (MCID) for the TDI.
Time Frame: Week 24 (Day 168)
Population: mITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 80 | 176
Scores on a scale | 1.6 (0.26) | 2.5 (0.17)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 mcg; UMEC versus Placebo; Test type: Other; p = 0.004, MMRM — Analysis performed using a MMRM model with covariates of treatment, BDI focal score, smoking status, country, Day, Day by BDI focal score and Day by treatment interactions; Least square Mean difference = 0.9, 95% CI 2-sided [0.3 to 1.5]

3. Secondary Outcome: Change From Baseline in Weighted Mean FEV1 Over 0 to 6 Hours Post-dose on Day 1
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Weighted mean FEV1 was calculated over the nominal 0 to 6 hour post dose period. Values from post-dose assessments which were actually before the time of dosing were excluded from the calculation. The 0 hour value is the average value obtained 30 minutes and 5 minutes pre-dose, and both the 0 hour and 6 hour values must be present for a 0- to 6 hour weighted mean to be calculated. The 0 -to 6 hour weighted mean was derived by calculating the area under the FEV1 curve over the nominal time points of 0 hour, 15 and 30 minutes, 1, 3 and 6 hours, using the trapezoidal rule, and then dividing by the actual time between dosing and the 6 hour assessment. Baseline value for FEV1 was calculated from the values measured 30 minutes and 5 minutes pre-dose on Day 1. Change from Baseline was calculated by subtracting the value on-treatment from the Baseline value.
Time Frame: Baseline (pre-dose on Day 1) and Day 1 (0 to 6 hours)
Population: mITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 203
Liters | 0.011 (0.0091) | 0.136 (0.0064)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 mcg; UMEC versus Placebo; Test type: Other; p < 0.001, ANCOVA — Analysis performed using an analysis of covariance (ANCOVA) model with covariates of treatment, baseline (mean of the two assessments made 30 min and 5 min pre-dose on Day 1), smoking status and country; Least square Mean difference = 0.125, 95% CI 2-sided [0.103 to 0.147]

4. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious AE (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or is associated with liver injury and impaired liver function.
Time Frame: Up to Day 178
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Participants
  AE | 56 | 122
  SAE | 9 | 17

5. Secondary Outcome: Change From Baseline in Vital Sign Parameters: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs (SBP and DBP) were obtained after participants had rested for approximately 5 minutes and before performing electrocardiogram (ECG) and spirometry testing. A single set of values was obtained. Baseline was the most recent recorded value before dosing on Day 1 at schedule visit. Change from Baseline was calculated by subtracting the value on-treatment from the Baseline value. Anytime post-Baseline values have been presented for SBP and DBP respectively.
Time Frame: Baseline (Day 1) to Day 169 (Visit 9)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Millimeters of mercury
  SBP, Anytime post-Baseline | 11.1 (11.25) | 11.4 (10.64)
  DBP, Anytime post-Baseline | -10.2 (7.55) | -10.8 (8.03)

6. Secondary Outcome: Change From Baseline in Vital Sign Parameter: Pulse Rate
Description: Vital sign pulse rate was obtained after participants had rested for approximately 5 minutes and before performing electrocardiogram (ECG) and spirometry testing. A single set of values was obtained. Baseline was the most recent recorded value before dosing on Day 1 at schedule visit. Change from Baseline was calculated by subtracting the value on-treatment from the Baseline value. Anytime post-Baseline values have been presented for pulse rate.
Time Frame: Baseline (Day 1) to Day 169 (Visit 9)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Beats/minute | 10.7 (10.94) | 8.2 (9.47)

7. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Any Time Post Baseline
Description: A 12-lead ECG measurement was obtained after measurement of vital signs and before spirometry testing. Participants should be placed in the supine position for the ECG measurements. Any ECG abnormality recorded by a participant after the start of study treatment was included in the any-time post-Baseline record of all ECG abnormalities. Partcipants with abnormal ECG interpretation have been presented.
Time Frame: Up to Day 169 (Visit 9)
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Participants | 51 | 105

8. Secondary Outcome: Number of Participants With Hematology Data Outside the Normal Range at Any Time Post-Baseline
Description: Hematology parameters included basophils (normal range 0 to 0.2 giga cells/Liter), eosinophils (0.05 to 0.55 giga cells/Liter), hematocrit (0.36 to 0.49 percentage of red blood cells in blood), hemoglobin (118 to 168 gram/Liter), lymphocytes (0.85 to 4.1 giga cells/Liter), monocytes (0.2 to 1.1 giga cells/Liter), platelet count (PC)(130 to 400 giga cells/Liter), neutrophils (1.8 to 8 giga cells/Liter), total neutrophils (TN) (1.8 to 8 giga cells/Liter), white blood cell [WBC] count (3.8 to 10.8 giga cells/Liter). Only categories with non-zero (high and low) values at any time post Baseline have been presented.
Time Frame: Up to Day 168 (Visit 8)
Population: mITT Population. Only those participants available at the specified time point were analyzed represented by n=x, x in the category titles.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 96 | 196
Participants
  Eosinophils, Any time post Baseline, High,n=96,196 | 8 | 11
  Eosinophils, Any time post Baseline, Low,n=96,196 | 19 | 37
  Hematocrit, Any time post Baseline, High,n=96,196 | 14 | 35
  Hematocrit, Any time post Baseline, Low,n=96,196 | 3 | 21
  Hemoglobin, Any time post Baseline, High,n=96,196 | 2 | 5
  Hemoglobin, Any time post Baseline, Low,n=96,196 | 7 | 28
  Lymphocytes, Any time post Baseline, High,n=96,196 | 1 | 3
  Lymphocytes, Any time post Baseline, Low,n=96,196 | 3 | 10
  Monocytes, Any time post Baseline, High,n=96,196 | 0 | 1
  Monocytes, Any time post Baseline, Low,n=96,196 | 14 | 28
  PC, Any time post Baseline, High, n=96,195: number analyzed (Participants) | 96 | 195
  PC, Any time post Baseline, High, n=96,195 | 1 | 0
  PC, Any time post Baseline, Low, n=96,195: number analyzed (Participants) | 96 | 195
  PC, Any time post Baseline, Low, n=96,195 | 7 | 15
  Neutrophils, Any time post Baseline, High,n=96,196 | 8 | 12
  Neutrophils,Any time post Baseline, Low,n=96,196 | 0 | 2
  TN, Any time post Baseline, High, n=96,196 | 8 | 12
  TN, Any time post Baseline, Low, n=96,196 | 0 | 2
  WBC count, Any time post Baseline, High,n=96,196 | 7 | 12
  WBC count, Any time post Baseline, Low,n=96,196 | 0 | 1

9. Secondary Outcome: Number of Participants With Clinical Chemistry Data Outside the Normal Range at Any Time Post-Baseline
Description: Clinical chemistry parameters assessed included albumin (normal range 32 to 50 grams/Liter [G/L]), alkaline phosphatase (20 to 125 international units/Liter [IU/L]), alanine aminotransferase [ALT] (0 to 48 IU/L), aspartate aminotransferase [AST] (0 to 55 IU/L), direct bilirubin (0 to 6 micromoles/liter [umol/l]), indirect bilirubin (0 to 22 umol/l), total bilirubin (0 to 22 umol/l), calcium (2.12 to 2.56 milimoles/liter [mmol/l]), chloride (95 to 108 mmol/l), carbon dioxide [CO2] content/bicarbonate (20 to 32 mmol/l), creatinine (67.2 to 129.1 umol/l), creatinine phosphokinase [CPK] (0 to 235 IU/L), gamma glutamyl transferase [GGT] (0 to75 IU/L), glucose (3.9 to 6.9 mmol/l), phosphorus (0.7 to 1.4 mmol/l), potassium (3.5 to 5.3 mmol/l), protein total (58 to 81 G/L), sodium (135 to 146 mmol/l), urea nitrogen (2.5 to 10.5 mmol/l), uric acid (240 to 510 umol/l). Only categories with non-zero (high and low) values at any time post Baseline have been presented.
Time Frame: Up to Day 168 (Visit 8)
Population: mITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 96 | 196
Participants
  ALT, Any time post Baseline, High | 5 | 5
  Albumin, Any time post Baseline, High | 0 | 1
  Albumin, Any time post Baseline, Low | 0 | 1
  Alkaline Phosphatase, Any time post Baseline, High | 3 | 5
  Alkaline Phosphatase, Any time post Baseline, Low | 0 | 1
  AST, Any time post Baseline, High | 0 | 3
  Calcium, Any time post Baseline, Low | 2 | 1
  CO2 content,Any time post Baseline, Low | 6 | 26
  Chloride, Any time post Baseline, High | 0 | 8
  Chloride, Any time post Baseline, Low | 2 | 2
  Creatine Kinase, Any time post Baseline, High | 4 | 4
  Creatinine, Any time post Baseline, High | 0 | 1
  Creatinine, Any time post Baseline, Low | 20 | 51
  Direct Bilirubin, Any time post Baseline, High | 1 | 4
  GGT, Any time post Baseline, High | 10 | 12
  Glucose, Any time post Baseline, High | 23 | 46
  Glucose, Any time post Baseline, Low | 2 | 1
  Indirect Bilirubin, Any time post Baseline, High | 2 | 5
  Phosphorus, Any time post Baseline, High | 9 | 8
  Phosphorus, Any time post Baseline, Low | 3 | 5
  Potassium, Any time post Baseline, High | 1 | 1
  Potassium, Any time post Baseline, Low | 4 | 4
  Sodium, Any time post Baseline, High | 1 | 1
  Sodium, Any time post Baseline, Low | 1 | 4
  Total Bilirubin, Any time post Baseline, High | 4 | 8
  Total Protein, Any time post Baseline, High | 1 | 2
  Total Protein, Any time post Baseline, Low | 0 | 1
  Urea nitrogen, Any time post Baseline, High | 5 | 5
  Urea nitrogen, Any time post Baseline, Low | 2 | 1
  Uric acid, Any time post Baseline, High | 6 | 13
  Uric acid, Any time post Baseline, Low | 13 | 10

10. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameters by Dipstick Method
Description: Urinalysis parameters assessed were urine ketones, urine bilirubin, urine glucose, urine leukocyte esterase test for detecting WBC and urine protein. In this dipstick test, the level of bilirubin, glucose, leukocyte esterase and protein in urine samples was recorded as negative, trace, 1+, 2+, and 3+ (the plus sign increases with a higher level of bilirubin, glucose, leukocyte esterase, or proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive). Urine samples were collected for the measurement of urinalysis parameters by dipstick method up to Day 168 (Visit 8). Only categories with significant values have been presented. Only those participants with data available at the indicated time point were analyzed.
Time Frame: Up to Day 168 (Visit 8)
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 80 | 178
Participants
  Urine Bilirubin, Day 168, 1+ | 2 | 2
  Urine Bilirubin, Day 168, 2+ | 1 | 0
  Urine Glucose, Day 168, 1+ | 3 | 6
  Urine Glucose, Day 168, 2+ | 2 | 1
  Urine Glucose, Day 168, 3+ | 2 | 2
  Urine Glucose, Day 168, Trace | 2 | 2
  Urine leukocyte esterase, Day 168, 1+ | 1 | 1
  Urine leukocyte esterase, Day 168, 2+ | 0 | 2
  Urine leukocyte esterase, Day 168, Trace | 4 | 2
  Urine protein, Day 168, 1+ | 2 | 1
  Urine protein, Day 168, 2+ | 1 | 0
  Urine protein, Day 168, Trace | 10 | 6

11. Secondary Outcome: Mean Urine Potential of Hydrogen (pH)
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 to 6.0). Urine samples were collected for the measurement of urine pH up to Day 168 (Visit 8). Only categories with significant values have been presented. Only those participants with data available at the indicated time point were analyzed.
Time Frame: Day 168 (Visit 8)
Population: mITT Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 80 | 178
pH | 6.16 (0.520) | 6.25 (0.632)

12. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Days 28, 84 and 168
Description: The SGRQ is designed to measure health-related quality of life (HRQoL) in participants with diseases of airway obstruction with the use of 76 items grouped into three domains: symptoms, activity and impact. The questions are designed to be self-completed by the participant based on recall of the past 4 weeks. Domain score =sum of the weighted scores for the non-missing items within each domain/maximum possible score for those non-missing items x 100. The SGRQ total score= sum of the weighted scores from all 76 items /maximum possible score for the SGRQ x100. Scores range from 0, representing the best possible health status, to 100, representing the worst possible health status. A decrease in score indicates an improvement in HRQoL whereas increase indicates deterioration in HRQoL. Baseline was the most recent recorded value before dosing on Day 1 at schedule visit. Change from Baseline was calculated by subtracting the value on-treatment from the Baseline value.
Time Frame: Baseline (Day 1) and Day 28, Day 84 and Day 168
Population: mITT Population. Only those participants available at the specified time points were analyzed (represented by n=x,x in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Scores on a scale
  Day 28, n=91,188: number analyzed (Participants) | 91 | 188
  Day 28, n=91,188 | -1.45 (1.174) | -5.84 (0.813)
  Day 84, n= 84,183: number analyzed (Participants) | 84 | 183
  Day 84, n= 84,183 | -2.46 (1.268) | -7.05 (0.860)
  Day 168, n=78,176: number analyzed (Participants) | 78 | 176
  Day 168, n=78,176 | -4.31 (1.316) | -7.34 (0.882)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 mcg; Day 28, UMEC Vs Placebo; Test type: Other; p = 0.002, MMRM — Analysis performed using a repeated measures model with covariates of treatment, Baseline (score prior to dosing on Day 1), smoking status, country, Day, Day by Baseline and Day by treatment interactions; Least sqaure mean difference = -4.39, 95% CI 2-sided [-7.21 to -1.58]
Statistical Analysis 2: Comparison: Placebo vs UMEC 62.5 mcg; Day 84, UMEC Vs Placebo; Test type: Other; p = 0.003, MMRM — [p-value comment as in outcome 12, analysis 1]; Least square mean difference = -4.59, 95% CI 2-sided [-7.61 to -1.57]
Statistical Analysis 3: Comparison: Placebo vs UMEC 62.5 mcg; Day 168, UMEC Vs Placebo; Test type: Other; p = 0.058, MMRM — [p-value comment as in outcome 12, analysis 1]; Least sqaure mean difference = -3.03, 95% CI 2-sided [-6.15 to 0.10]

13. Secondary Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) Score at Days 28, 84 and 168
Description: The CAT is an 8-item, participant-completed instrument that covers symptoms such as cough, phlegm, chest tightness and breathlessness, and disease impacts including physical activity, confidence, sleep and energy. The CAT asks participant to score each item according to their current experience; there is no specific recall period. Items are scored on a 6-point response scale, with a score of 0 representing the participants are not experiencing the symptom/impact at all and a score of 5 representing a maximal symptom or impact. All items have equal weighting and so the total score is simply the sum of all scores and can range from 0 to a maximum of 40, with higher scores indicating a worse health state while a decrease in score indicates an improvement in health status. Baseline was the most recent recorded value before dosing on Day 1 at schedule visit. Change from Baseline was calculated by subtracting the value on-treatment from the Baseline value.
Time Frame: Baseline (Day 1) and Days 28, 84 and 168
Population: mITT Population. Only those participants available at the specified time points were analyzed (represented by n=x, x in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Scores on a scale
  Day 28, n=94,199: number analyzed (Participants) | 94 | 199
  Day 28, n=94,199 | -0.26 (0.551) | -1.75 (0.378)
  Day 84, n=87,189: number analyzed (Participants) | 87 | 189
  Day 84, n=87,189 | -0.08 (0.594) | -2.18 (0.403)
  Day 168, n=80,179: number analyzed (Participants) | 80 | 179
  Day 168, n=80,179 | -1.32 (0.648) | -2.00 (0.434)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 mcg; Day 28, UMEC Vs Placebo; Test type: Other; p = 0.027, MMRM — [p-value comment as in outcome 12, analysis 1]; Least sqaure mean difference = -1.49, 95% CI 2-sided [-2.81 to -0.17]
Statistical Analysis 2: Comparison: Placebo vs UMEC 62.5 mcg; Day 84, UMEC Vs Placebo; Test type: Other; p = 0.004, MMRM — [p-value comment as in outcome 12, analysis 1]; Least square mean difference = -2.10, 95% CI 2-sided [-3.51 to -0.68]
Statistical Analysis 3: Comparison: Placebo vs UMEC 62.5 mcg; Day 128, UMEC Vs Placebo; Test type: Other; p = 0.386, MMRM — [p-value comment as in outcome 12, analysis 1]; Least square mean difference = -0.68, 95% CI 2-sided [-2.22 to 0.86]

14. Secondary Outcome: Number of Participants With Healthcare Resource Utilization Status
Description: The total number of participants with visits for each type of healthcare contact ( office/practice visits, urgent care/outpatient clinic visits, emergency room visits and the intensive care visit and general wards visit have been presented.
Time Frame: Up to Day 169 (Visit 9)
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Participants
  Office/Practice Visits | 4 | 12
  Urgent Care/Outpatient Clinic Visits | 11 | 10
  Emergency Room Visits | 1 | 1

15. Secondary Outcome: Number of Days Requiring Admission to Intensive Care Unit and General Ward
Description: The total number of days requiring admission to intensive care unit and general ward have been presented.
Time Frame: Up to Day 169 (Visit 9)
Population: mITT Population
Measure: Number; unit: Days
Arm/Group | Placebo | UMEC 62.5 mcg
Number analyzed (Participants) | 101 | 205
Days
  Days in Intensive Care Unit | 0 | 0
  Days in General Ward | 35 | 20

ADVERSE EVENTS:
Time Frame: AE and nSAE were collected from Day 1 to Day 178
Description: mITT population was used to assess AE and nSAE.
Arm/Group | Placebo | UMEC 62.5 mcg
All-Cause Mortality (participants affected / at risk) | 0/101 | 1/205
Serious Adverse Events (participants affected / at risk) | 9/101 | 17/205
Other Adverse Events (participants affected / at risk) | 32/101 | 52/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=101) | UMEC 62.5 mcg (N=205)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pneumonia (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Chest pain (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=101) | UMEC 62.5 mcg (N=205)
Upper respiratory tract infection (Infections and infestations) | 13 | 25
Nasopharyngitis (Infections and infestations) | 11 | 19
Urinary tract infection (Infections and infestations) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 6
Blood glucose increased (Investigations) | 3 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT02184611/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT02184611/SAP_001.pdf